CLINICAL TRIAL: NCT06418633
Title: Variations in the Hemostatic System Induced by a Standardized Walking Test: Controls Vs. Cases with a History of Non-anticoagulated Venous Thromboembolic Disease
Brief Title: Variations in the Hemostatic System Induced by a Standardized Walking Test
Acronym: FAST&THROMBIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIMAO 2023 1
Record Dates: First submitted 2024-04-28; First posted 2024-05-17 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Venous Thromboembolism
Keywords: Physical exercise
MeSH Terms: conditions — Venous Thromboembolism; Motor Activity | interventions — Blood Pressure Monitors

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, cross-sectional, proof-of-concept study,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (Active Comparator): Subjects with neither a personal history nor family history of venous thromboembolism in first-degree relatives.
  Interventions: Other: 60-minute walking test; Diagnostic Test: Static blood test; Diagnostic Test: Post-effort blood test; Other: Electrocardiogram; Other: Blood pressure monitoring
- Patients (Active Comparator): Patients with a personal history of induced venous thromboembolism, the last attack dating back to more than 6 months, whose clinical phenotype did not justify long-term antithrombotic drug prophylaxis
  Interventions: Other: 60-minute walking test; Diagnostic Test: Static blood test; Diagnostic Test: Post-effort blood test; Other: Electrocardiogram; Other: Blood pressure monitoring
- Individual reproducibility" subgroup: controls (Active Comparator): 10 subjects with neither a personal history nor family history of venous thromboembolism in first-degree relatives who have accepted to re-do the test one week later.
  Interventions: Other: 60-minute walking test; Diagnostic Test: Static blood test; Diagnostic Test: Post-effort blood test; Other: Electrocardiogram; Other: Blood pressure monitoring
- Individual reproducibility" subgroup: patients (Active Comparator): 10 patients with a history of induced venous thromboembolism, the last attack dating back to more than 6 months, whose clinical phenotype did not justify long-term antithrombotic drug prophylaxis, who have accepted to re-do the test one week later.
  Interventions: Other: 60-minute walking test; Diagnostic Test: Static blood test; Diagnostic Test: Post-effort blood test; Other: Electrocardiogram; Other: Blood pressure monitoring

INTERVENTIONS:
Other: 60-minute walking test — Treadmill walking test in the morning, 2 hours after breakfast, following a clinical examination, resting 12-lead electrocardiogram and blood pressure measurement. After a 3-minute warm-up and walking of speed 2.5 km per hour, no incline, the speed and incline are gradually increased to reach a target heart rate close to the theoretical ventilatory threshold, around 70% of the theoretical maximum value (evaluated by Astrand's formula: 220-age), i.e. aerobic conditions of moderate intensity so that prolonged effort can be maintained. Test performed in presence of a physician trained in stress testing. Emergency cart and defibrillator available in the department. Intra-hospital vital emergency protocol in place, with resuscitation teams on standby. The cardiology department, in the same building, can be contacted in the event of a cardiological abnormality during the test or recovery. The test takes 60 minutes, including a 3-minute initial warm-up.
Diagnostic Test: Static blood test — 33.3 ml of blood will be taken from each participant whilst at rest, before undergoing the 60-minute walking test
Diagnostic Test: Post-effort blood test — 33.3 ml of blood will be taken from each participant immediately after undergoing the 60-minute walking test.
Other: Electrocardiogram — An electrocardiogram will be carried out throughout the exercise period and during the first 30 minutes of recovery.
Other: Blood pressure monitoring — Blood pressure will be monitored out throughout the exercise period and during the first 30 minutes of recovery.

SUMMARY:
Two groups of patients will be compared: One group of patients with a history of venous thromboembolic disease and one group without. Both groups will be subjected to a walking test and with electrocardiogram measurements and blood tests.

DETAILED DESCRIPTION:
Induced venous thromboembolism is a situation in which venous thromboembolic disease is triggered by an acute event that activates hemostasis: surgery, trauma, infectious or inflammatory outbreak, etc., a situation in which the risk of spontaneous recurrence, in the absence of a new provoking circumstance, is low, leading to the suggestion, not of long-term thromboprophylaxis, but simply the transient prevention of an event when there is a new clinical event likely to activate hemostasis. One such event is acute physical exertion.

Indeed, cohort studies seem to show that regular physical activity is associated with a low incidence of venous thromboembolism. Trained individuals have an endogenous thrombotic potential, assessed by the thrombin TGT test, lower than that of sedentary controls. A 3-month regimen of daily endurance exercise reduces thrombin generation controls and optimizes the fibrinolytic system. Repetitive exercise is accompanied by a depletion of exercise-induced platelet activation. However, several cases of venous thromboembolism have been reported in high-level athletes without usual risk factors and acute high-intensity rowing induces an acute increase in thrombin generation immediately after exercise, which disappears within 16 to 24 hours. The relationship between the level of physical activity and the risk of VTE could be a U-shaped relation, with an increasing risk of event in intense acute practice.

However, no data exists on the hemostatic impact of an acute session of physical activity in patients with a history of venous thromboembolism. Thus, the hypothesis is that exercise-induced response of hemostasis differ in patients with an history of provoked VTE compared to subjects without a history of venous thromboembolism.

This is a proof-of-concept, pathophysiological, single-center, cross-sectional, prospective comparison study of a group of patients with a personal history of induced Venous thromboembolism to a group of sex- and age- and sex-matched controls (+/- 5 years).

- Type of clinical study: Stress test-induced variations in parameters describing the results of the thrombin generation test (Thromboscreen®) in a group of Patients (Cases) will be compared with those obtained in a group of Control subjects (Controls) with a ratio 1:1.

The Patients group comprises 47 patients with a personal history of induced venous thromboembolism, the last event dating back to more than 6 months, whose clinical phenotype did not justify long-term antithrombotic drug prophylaxis.The Control group comprises 47 patients with no personal history of venous thromboembolism and no family history of venous thromboembolism in first-degree relatives.

The study intervention consists of an hour-long walking test and two blood tests in both groups for all participants (Controls and Patients).

- Intra-individual reproducibility will be analyzed in 20 subjects (10 patients and 10 controls) who will take the walking test twice on two separate days.

Patients will be selected during a venous thromboembolism follow-up consultation by a physician from either department (Vascular Medicine Consultation or Biological Hematology and Consultations).Inclusion and non-inclusion criteria will be checked, and the study will be explained to participants (patients and controls).Patients and controls will be systematically asked to take part in the variability analysis on a voluntary basis, until 10 subjects per group have agreed to carry out the second test.

The walking test is performed in the morning, 2 hours after a standard breakfast, on a treadmill. It will be preceded by a clinical examination, a resting 12-lead electrocardiogram and a brachial pressure measurement. After a 3-minute warm-up and "habituation" period (walking speed 2.5 km per hour with no incline), the speed and incline will be gradually increased until a target heart rate close to the theoretical ventilatory threshold, and of the order of 70% of the theoretical maximum value (evaluated by Astrand's formula: 220-age), so as to maintain aerobic exercise conditions of moderate intensity, enabling prolonged effort to be maintained. Blood samples will be taken from each participant whilst at rest, before undergoing the 60-minute walking test, in a sitting position, and just after the exercise test.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria common to both groups :
* Patients who have given written informed consent.
* Patients who are affiliated to or beneficiaries of a social security scheme.

Inclusion criteria specific to the Patient Group:

* Patients with a personal history of provoked venous thromboembolism, venous thrombosis and/or pulmonary embolism, with the last attack dating back to more than 6 months, and whose clinical phenotype did not justify long-term antithrombotic drug prophylaxis.

Definition of provoked venous thromboembolism : The clinical criteria used to classify venous thromboembolism as provoked are :

* First year of combined oestrogen-progestogen oral contraception, or contraception using an oestrogen-impregnated vaginal ring or transcutaneous synthetic oestrogen patch.
* Hormonal stimulation for oocyte retrieval
* Pregnancy and 6 weeks post-partum
* Surgery
* Trauma
* Immobilisation in plaster or splint
* Outbreak of acute infectious disease
* Acute flare-up of inflammatory disease
* Prolonged air travel lasting at least 4 hours
* Prolonged strict bed rest lasting at least 3 consecutive days.

Inclusion criteria specific to the Control Group:

* Subjects with no personal history of venous thromboembolism
* Subjects with no family history of venous thromboembolism in first-degree relatives
* Subjects of the same sex and age with a tolerance of +/- 5 years in relation to the matched case.

Exclusion Criteria:

* Patients who are physically unable to perform the 60-minute walking test, for any reason, in particular cardiovascular contraindications to exercise (recent acute coronary syndrome unstable angina, rhythm disorders, tight aortic stenosis, cardiac heart failure, acute myocarditis, pericarditis or endocarditis endocarditis, poorly controlled hypertension, pre-stress blood pressure > 200/110 mmHg, recent stroke or transient ischemic attack).
* Patients on anticoagulant or antithrombotic treatment, ongoing or discontinued within the last month.
* Patients treated for pulmonary embolism who remain dyspneic after anticoagulant treatment and requiring a work-up for pulmonary hypertension.
* Last surgery dating back to less than 3 months.
* Known chronic morbidities: diabetes mellitus, chronic inflammatory or infectious disease, heart failure, renal insufficiency, hepatic insufficiency or arterial thrombosis dating back to less than 3 months.
* For women: treatment containing synthetic or natural estrogen, in progress or discontinued for less than a month
* Pregnancy within the last year.
* Difficult venous access.
* Regular practice of an intensive sporting/physical activity, such as running, tennis, cycling etc. of more than 3 hours per week.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Thrombin generation dosage before effort in controls | Day 0
  The amount of thrombomodulin in the blood will be measured in nmol/L with the help of Thromboscreen(TM)
Thrombin generation dosage before effort in patients | Day 0
  The amount of thrombomodulin in the blood will be measured in nmol/L with the help of Thromboscreen(TM)
Thrombin generation dosage after effort in controls | Day 0
  The amount of thrombomodulin in the blood will be measured in nmol/L with the help of Thromboscreen(TM). The difference between measurements before and after effort will be measured in nM.min-1
Thrombin generation dosage after effort in patients | Day 0
  The amount of thrombomodulin in the blood will be measured in nmol/L with the help of Thromboscreen(TM). The difference between measurements before and after effort will be measured in nM.min-1
Thrombin generation dosage before effort in the "Individual reproducibility" subgroup: controls | Day 7
  The amount of thrombomodulin in the blood will be measured in nmol/L with the help of Thromboscreen(TM)
Thrombin generation dosage before effort in the "Individual reproducibility" subgroup: patients | Day 7
  The amount of thrombomodulin in the blood will be measured in nmol/L with the help of Thromboscreen(TM)
Thrombin generation dosage after effort in the "Individual reproducibility" subgroup: controls | Day 7
  The amount of thrombomodulin in the blood will be measured in nmol/L with the help of Thromboscreen(TM). The difference between measurements before and after effort will be measured in nM.min-1
Thrombin generation dosage after effort in the "Individual reproducibility" subgroup: patients | Day 7
  The amount of thrombomodulin in the blood will be measured in nmol/L with the help of Thromboscreen(TM). The difference between measurements before and after effort will be measured in nM.min-1

SECONDARY OUTCOMES:
Distribution in the Control group | Day 0
  Measurements in nM.min-1 will be compared to elicit central tendency, dispersion and heterogeneity in the Control group
Distribution in the Patient group | Day 0
  Measurements in nM.min-1 will be compared to elicit central tendency, dispersion and heterogeneity in the Patient group
Thromboscreen test in Controls in the absence of thrombomodulin : Latency time | Day 0
  Latency time in the absence of thrombomodulin will be measured in seconds in Controls.
Thromboscreen test in Controls in the absence of thrombomodulin : Thrombin peak intensity | Day 0
  Thrombin peak intensity in the absence of thrombomodulin will be measured in Controls.
Thromboscreen test in Controls in the absence of thrombomodulin : Time-to-peak thrombin | Day 0
  Time-to-peak thrombin in the absence of thrombomodulin will be measured in Controls.
Thromboscreen test in Controls in the absence of thrombomodulin : Initial thrombin generation velocity | Day 0
  Initial thrombin generation velocity in the absence of thrombomodulin will be measured in seconds in Controls.
Thromboscreen test in Controls in the absence of thrombomodulin : Time to return to baseline | Day 0
  Time to return to baseline in the absence of thrombomodulin will be measured in seconds in Controls.
Thromboscreen test in Controls in the presence of thrombomodulin : Latency time | Day 0
  Latency time in the presence of thrombomodulin will be measured in seconds in Controls.
Thromboscreen test in Controls in the presence of thrombomodulin : Thrombin peak intensity | Day 0
  Thrombin peak intensity in the presence of thrombomodulin will be measured in Controls.
Thromboscreen test in Controls in the presence of thrombomodulin : Time-to-peak thrombin | Day 0
  Time-to-peak thrombin in the presence of thrombomodulin will be measured in Controls.
Thromboscreen test in Controls in the presence of thrombomodulin : Initial thrombin generation velocity | Day 0
  Initial thrombin generation velocity in the presence of thrombomodulin will be measured in seconds in Controls.
Thromboscreen test in Controls in the presence of thrombomodulin : Time to return to baseline | Day 0
  Time to return to baseline in the presence of thrombomodulin will be measured in seconds in Controls.
Thromboscreen test in Patients in the absence of thrombomodulin : Latency time | Day 0
  Latency time in the absence of thrombomodulin will be measured in seconds in Patients.
Thromboscreen test in Patients in the absence of thrombomodulin : Thrombin peak intensity | Day 0
  Thrombin peak intensity in the absence of thrombomodulin will be measured in Patients.
Thromboscreen test in Patients in the absence of thrombomodulin : Time-to-peak thrombin | Day 0
  Time-to-peak thrombin, initial thrombin generation velocity, time to return to baseline for the thrombin generation test performed in the absence of thrombomodulin will be measured in seconds in Patients.
Thromboscreen test in Patients in the absence of thrombomodulin : Initial thrombin generation velocity | Day 0
  Initial thrombin generation velocity in the absence of thrombomodulin will be measured in seconds in Patients.
Thromboscreen test in Patients in the absence of thrombomodulin : Time to return to baseline | Day 0
  Time to return to baseline in the absence of thrombomodulin will be measured in seconds in Patients.
Thromboscreen test in Patients in the presence of thrombomodulin : Latency time | Day 0
  Latency time in the presence of thrombomodulin will be measured in seconds in Patients.
Thromboscreen test in Patients in the presence of thrombomodulin : Thrombin peak intensity | Day 0
  Thrombin peak intensity in the presence of thrombomodulin will be measured in seconds in Patients.
Thromboscreen test in Patients in the presence of thrombomodulin : Time-to-peak thrombin | Day 0
  Time-to-peak thrombin in the presence of thrombomodulin be measured in seconds in Patients.
Thromboscreen test in Patients in the presence of thrombomodulin : Initial thrombin generation velocity | Day 0
  Initial thrombin generation velocity in the presence of thrombomodulin will be measured in seconds in Patients.
Thromboscreen test in Patients in the presence of thrombomodulin : Time to return to baseline | Day 0
  Time to return to baseline in the presence of thrombomodulin will be measured in seconds in Patients.
Distribution of other parameters of the Thromboscreen test in Controls | Day 0
  The distribution (central tendency, dispersion, heterogeneity), of the various biological parameters (latency time, thrombin peak intensity, time-to-peak thrombin, initial thrombin generation velocity, time to return to baseline) will be measured in Controls
Distribution of other parameters of the Thromboscreen test in Patients | Day 0
  The distribution (central tendency, dispersion, heterogeneity), of the various biological parameters (latency time, thrombin peak intensity, time-to-peak thrombin, initial thrombin generation velocity, time to return to baseline) will be measured in Patients
Endogenous Thrombotic Potential in the presence of thrombomodulin in Controls | Day 0
  nM.min
Endogenous Thrombotic Potential in the absence of thrombomodulin in Controls | Day 0
  nM.min
Endogenous Thrombotic Potential in the presence of thrombomodulin in Patients | Day 0
  nM.min
Endogenous Thrombotic Potential in the absence of thrombomodulin in Patients | Day 0
  nM.min
Heterogeneity of Endogenous Thrombotic Potential in Controls | Day 0
  Statistical analysis, Cochrane's Q test
Heterogeneity of Endogenous Thrombotic Potential in Patients | Day 0
  Statistical analysis, Cochrane's Q test
Complete Blood Count in Controls before the walking test: White blood cells | Day 0
  White blood cells will be measured in thousands/µL
Complete Blood Count in Controls before the walking test: White blood cells | Day 7
  White blood cells will be measured in thousands/µL
Complete Blood Count in Controls after the walking test: White blood cells | Day 0
  White blood cells will be measured in thousands/µL
Complete Blood Count in Controls after the walking test: White blood cells | Day 7
  White blood cells will be measured in thousands/µL
Complete Blood Count in Patients before the walking test: White blood cells | Day 0
  White blood cells will be measured in thousands/µL
Complete Blood Count in Patients before the walking test: White blood cells | Day 7
  White blood cells will be measured in thousands/µL
Complete Blood Count in Patients after the walking test: White blood cells | Day 0
  White blood cells will be measured in thousands/µL
Complete Blood Count in Patients after the walking test: White blood cells | Day 7
  White blood cells will be measured in thousands/µL
Complete Blood Count in Controls before the walking test: Red blood cells | Day 0
  Red blood cells will be measured in millions per cubic millimeter
Complete Blood Count in Controls before the walking test: Red blood cells | Day 7
  Red blood cells will be measured in millions per cubic millimeter
Complete Blood Count in Patients before the walking test: Red blood cells | Day 0
  Red blood cells will be measured in millions per cubic millimeter
Complete Blood Count in Patients before the walking test: Red blood cells | Day 7
  Red blood cells will be measured in millions per cubic millimeter
Complete Blood Count in Controls after the walking test: Red blood cells | Day 0
  Red blood cells will be measured in millions per cubic millimeter
Complete Blood Count in Controls after the walking test: Red blood cells | Day 7
  Red blood cells will be measured in millions per cubic millimeter
Complete Blood Count in Patients after the walking test: Red blood cells | Day 0
  Red blood cells will be measured in millions per cubic millimeter
Complete Blood Count in Patients after the walking test: Red blood cells | Day 7
  Red blood cells will be measured in millions per cubic millimeter
Complete Blood Count in Controls before the walking test:Hemaglobin | Day 0
  Hemaglobin will be measured in g/L
Complete Blood Count in Controls before the walking test:Hemaglobin | Day 7
  Hemaglobin will be measured in g/L
Complete Blood Count in Patients before the walking test:Hemaglobin | Day 0
  Hemaglobin will be measured in g/L
Complete Blood Count in Patients before the walking test:Hemaglobin | Day 7
  Hemaglobin will be measured in g/L
Complete Blood Count in Controls after the walking test: Hemaglobin | Day 0
  Hemaglobin will be measured in g/L
Complete Blood Count in Controls after the walking test: Hemaglobin | Day 7
  Hemaglobin will be measured in g/L
Complete Blood Count in Patients after the walking test: Hemaglobin | Day 0
  Hemaglobin will be measured in g/L
Complete Blood Count in Patients after the walking test: Hemaglobin | Day 7
  Hemaglobin will be measured in g/L
Complete Blood Count in Controls before the walking test: Hematocrite | Day 0
  Hematrocrite will be measured in L/L
Complete Blood Count in Controls before the walking test: Hematocrite | Day 7
  Hematrocrite will be measured in L/L
Complete Blood Count in Patients before the walking test: Hematocrite | Day 0
  Hematrocrite will be measured in L/L
Complete Blood Count in Patients before the walking test: Hematocrite | Day 7
  Hematrocrite will be measured in L/L
Complete Blood Count in Controls after the walking test: Hematocrite | Day 0
  Hematrocrite will be measured in L/L
Complete Blood Count in Controls after the walking test: Hematocrite | Day 7
  Hematrocrite will be measured in L/L
Complete Blood Count in Patients after the walking test: Hematocrite | Day 0
  Hematrocrite will be measured in L/L
Complete Blood Count in Patients after the walking test: Hematocrite | Day 7
  Hematrocrite will be measured in L/L
Complete Blood Count in Controls before the walking test: mean corpuscular volume | Day 0
  Mean corpuscular volume will be measured in fL
Complete Blood Count in Controls before the walking test: mean corpuscular volume | Day 7
  Mean corpuscular volume will be measured in fL
Complete Blood Count in Patients before the walking test: mean corpuscular volume | Day 0
  Mean corpuscular volume will be measured in fL
Complete Blood Count in Patients before the walking test: mean corpuscular volume | Day 7
  Mean corpuscular volume will be measured in fL
Complete Blood Count in Controls after the walking test: mean corpuscular volume | Day 0
  Mean corpuscular volume will be measured in fL
Complete Blood Count in Controls after the walking test: mean corpuscular volume | Day 7
  Mean corpuscular volume will be measured in fL
Complete Blood Count in Patients after the walking test: mean corpuscular volume | Day 0
  Mean corpuscular volume will be measured in fL
Complete Blood Count in Patients after the walking test: mean corpuscular volume | Day 7
  Mean corpuscular volume will be measured in fL
Complete Blood Count in Controls before the walking test: mean corpuscular hemoglobin | Day 0
  Mean Corpuscular Hemoglobin will be measured in pg
Complete Blood Count in Controls before the walking test: mean corpuscular hemoglobin | Day 7
  Mean Corpuscular Hemoglobin will be measured in pg
Complete Blood Count in Patients before the walking test: mean corpuscular hemoglobin | Day 0
  Mean Corpuscular Hemoglobin will be measured in pg
Complete Blood Count in Patients before the walking test: mean corpuscular hemoglobin | Day 7
  Mean Corpuscular Hemoglobin will be measured in pg
Complete Blood Count in Controls after the walking test: Mean corpuscular hemoglobin | Day 0
  Mean Corpuscular Hemoglobin will be measured in pg
Complete Blood Count in Controls after the walking test: Mean corpuscular hemoglobin | Day 7
  Mean Corpuscular Hemoglobin will be measured in pg
Complete Blood Count in Patients after the walking test: Mean corpuscular hemoglobin | Day 0
  Mean Corpuscular Hemoglobin will be measured in pg
Complete Blood Count in Patients after the walking test: Mean corpuscular hemoglobin | Day 7
  Mean Corpuscular Hemoglobin will be measured in pg
Complete Blood Count in Controls before the walking test: Mean corpuscular hemoglobin concentration | Day 0
  Mean Corpuscular Hemoglobin Concentration will be measured in g/L
Complete Blood Count in Controls before the walking test: Mean corpuscular hemoglobin concentration | Day 7
  Mean Corpuscular Hemoglobin Concentration will be measured in g/L
Complete Blood Count in Patients before the walking test: Mean corpuscular hemoglobin concentration | Day 0
  Mean Corpuscular Hemoglobin Concentration will be measured in g/L
Complete Blood Count in Patients before the walking test: Mean corpuscular hemoglobin concentration | Day 7
  Mean Corpuscular Hemoglobin Concentration will be measured in g/L
Complete Blood Count in Controls after the walking test: Mean corpuscular hemoglobin concentration | Day 0
  Mean Corpuscular Hemoglobin Concentration will be measured in g/L
Complete Blood Count in Controls after the walking test: Mean corpuscular hemoglobin concentration | Day 7
  Mean Corpuscular Hemoglobin Concentration will be measured in g/L
Complete Blood Count in Patients after the walking test: Mean corpuscular hemoglobin concentration | Day 0
  Mean Corpuscular Hemoglobin Concentration will be measured in g/L
Complete Blood Count in Patients after the walking test: Mean corpuscular hemoglobin concentration | Day 7
  Mean Corpuscular Hemoglobin Concentration will be measured in g/L
Complete Blood Count in Controls before the walking test: red cell distribution width | Day 0
  Red cell distribution width will be measured as %
Complete Blood Count in Controls before the walking test: red cell distribution width | Day 7
  Red cell distribution width will be measured as %
Complete Blood Count in Patients before the walking test: red cell distribution width | Day 0
  Red cell distribution width will be measured as %
Complete Blood Count in Patients before the walking test: red cell distribution width | Day 7
  Red cell distribution width will be measured as %
Complete Blood Count in Controls after the walking test: red cell distribution width | Day 0
  Red cell distribution width will be measured as %
Complete Blood Count in Controls after the walking test: red cell distribution width | Day 7
  Red cell distribution width will be measured as %
Complete Blood Count in Patients after the walking test: red cell distribution width | Day 0
  Red cell distribution width will be measured as %
Complete Blood Count in Patients after the walking test: red cell distribution width | Day 7
  Red cell distribution width will be measured as %
Complete Blood Count in Controls before the walking test: Platelets | Day 0
  Platelets will be measured in thousands/µL
Complete Blood Count in Controls before the walking test: Platelets | Day 7
  Platelets will be measured in thousands/µL
Complete Blood Count in Patients before the walking test: Platelets | Day 0
  Platelets will be measured in thousands/µL
Complete Blood Count in Patients before the walking test: Platelets | Day 7
  Platelets will be measured in thousands/µL
Complete Blood Count in Controls after the walking test: Platelets | Day 0
  Platelets will be measured in thousands/µL
Complete Blood Count in Controls after the walking test: Platelets | Day 7
  Platelets will be measured in thousands/µL
Complete Blood Count in Patients after the walking test: Platelets | Day 0
  Platelets will be measured in thousands/µL
Complete Blood Count in Patients after the walking test: Platelets | Day 7
  Platelets will be measured in thousands/µL
Complete Blood Count in Controls before the walking test: Neutrophils | Day 0
  Neutrophils will be measured in thousands/µL
Complete Blood Count in Controls before the walking test: Neutrophils | Day 7
  Neutrophils will be measured in thousands/µL
Complete Blood Count in Patients before the walking test: Neutrophils | Day 0
  Neutrophils will be measured in thousands/µL
Complete Blood Count in Patients before the walking test: Neutrophils | Day 7
  Neutrophils will be measured in thousands/µL
Complete Blood Count in Controls after the walking test: Neutrophils | Day 0
  Neutrophils will be measured in thousands/µL
Complete Blood Count in Controls after the walking test: Neutrophils | Day 7
  Neutrophils will be measured in thousands/µL
Complete Blood Count in Patients after the walking test: Neutrophils | Day 0
  Neutrophils will be measured in thousands/µL
Complete Blood Count in Patients after the walking test: Neutrophils | Day 7
  Neutrophils will be measured in thousands/µL
Complete Blood Count in Controls before the walking test: Lymphocytes | Day 0
  Lymphocytes will be measured in thousands/µL
Complete Blood Count in Controls before the walking test: Lymphocytes | Day 7
  Lymphocytes will be measured in thousands/µL
Complete Blood Count in Patients before the walking test: Lymphocytes | Day 0
  Lymphocytes will be measured in thousands/µL
Complete Blood Count in Patients before the walking test: Lymphocytes | Day 7
  Lymphocytes will be measured in thousands/µL
Complete Blood Count in Controls after the walking test: Lymphocytes | Day 0
  Lymphocytes will be measured in thousands/µL
Complete Blood Count in Controls after the walking test: Lymphocytes | Day 7
  Lymphocytes will be measured in thousands/µL
Complete Blood Count in Patients after the walking test: Lymphocytes | Day 0
  Lymphocytes will be measured in thousands/µL
Complete Blood Count in Patients after the walking test: Lymphocytes | Day 7
  Lymphocytes will be measured in thousands/µL
Complete Blood Count in Controls before the walking test: Monocytes | Day 0
  Monocytes will be measured in thousands/µL
Complete Blood Count in Controls before the walking test: Monocytes | Day 7
  Monocytes will be measured in thousands/µL
Complete Blood Count in Patients before the walking test: Monocytes | Day 0
  Monocytes will be measured in thousands/µL
Complete Blood Count in Patients before the walking test: Monocytes | Day 7
  Monocytes will be measured in thousands/µL
Complete Blood Count in Controls after the walking test: Monocytes | Day 0
  Monocytes will be measured in thousands/µL
Complete Blood Count in Controls after the walking test: Monocytes | Day 7
  Monocytes will be measured in thousands/µL
Complete Blood Count in Patients after the walking test: Monocytes | Day 0
  Monocytes will be measured in thousands/µL
Complete Blood Count in Patients after the walking test: Monocytes | Day 7
  Monocytes will be measured in thousands/µL
Complete Blood Count in Controls before the walking test: Eosinophils | Day 0
  Eosinophils will be measured in hundreds/µL
Complete Blood Count in Controls before the walking test: Eosinophils | Day 7
  Eosinophils will be measured in hundreds/µL
Complete Blood Count in Patients before the walking test: Eosinophils | Day 0
  Eosinophils will be measured in hundreds/µL
Complete Blood Count in Patients before the walking test: Eosinophils | Day 7
  Eosinophils will be measured in hundreds/µL
Complete Blood Count in Controls after the walking test: Eosinophils | Day 0
  Eosinophils will be measured in hundreds/µL
Complete Blood Count in Controls after the walking test: Eosinophils | Day 7
  Eosinophils will be measured in hundreds/µL
Complete Blood Count in Patients after the walking test: Eosinophils | Day 0
  Eosinophils will be measured in hundreds/µL
Complete Blood Count in Patients after the walking test: Eosinophils | Day 7
  Eosinophils will be measured in hundreds/µL
Complete Blood Count in Controls before the walking test: Basophils | Day 0
  Basophils will be measured in thousands/µL
Complete Blood Count in Controls before the walking test: Basophils | Day 7
  Basophils will be measured in thousands/µL
Complete Blood Count in Patients before the walking test: Basophils | Day 0
  Basophils will be measured in thousands/µL
Complete Blood Count in Patients before the walking test: Basophils | Day 7
  Basophils will be measured in thousands/µL
Complete Blood Count in Controls after the walking test: Basophils | Day 0
  Basophils will be measured in thousands/µL
Complete Blood Count in Controls after the walking test: Basophils | Day 7
  Basophils will be measured in thousands/µL
Complete Blood Count in Patients after the walking test: Basophils | Day 0
  Basophils will be measured in thousands/µL
Complete Blood Count in Patients after the walking test: Basophils | Day 7
  Basophils will be measured in thousands/µL
NETosis markers in Controls before the walking test | Day 0
  Fluorescence signal intensity of neutrophils will be measured on a SYSMEX automat
NETosis markers in Controls after the walking test | Day 0
  Fluorescence signal intensity of neutrophils will be measured on a SYSMEX automat
NETosis markers in Patients before the walking test | Day 7
  Fluorescence signal intensity of neutrophils will be measured on a SYSMEX automat
NETosis markers in Patients after the walking test | Day 7
  Fluorescence signal intensity of neutrophils will be measured on a SYSMEX automat
NETosis markers in Controls before the walking test: reacting monocytes | Day 0
  The percentage of reacting monocytes will be measured on a SYSMEX automat
NETosis markers in Controls after the walking test: reacting monocytes | Day 0
  The percentage of reacting monocytes will be measured on a SYSMEX automat
NETosis markers in Controls before the walking test: reacting monocytes | Day 7
  The percentage of reacting monocytes will be measured on a SYSMEX automat
NETosis markers in Controls after the walking test: reacting monocytes | Day 7
  The percentage of reacting monocytes will be measured on a SYSMEX automat
NETosis markers in Controls before the walking test: reacting lymphocytes | Day 0
  The percentage of reacting lymphocytes will be measured on a SYSMEX automat
NETosis markers in Controls after the walking test: reacting lymphocytes | Day 0
  The percentage of reacting lymphocytes will be measured on a SYSMEX automat
NETosis markers in Patients before the walking test: reacting lymphocytes | Day 7
  The percentage of reacting lymphocytes will be measured on a SYSMEX automat
NETosis markers in Patients after the walking test: reacting lymphocytes | Day 7
  The percentage of reacting lymphocytes will be measured on a SYSMEX automat
NETosis markers in Controls before the walking test: | Day 0
  The percentage of reacting lymphocytes will be measured on a SYSMEX automat
NETosis markers in Controls after the walking test: circulating citrulinated histone H3 | Day 0
  The percentage of circulating citrulinated histone H3 will be measured on a SYSMEX automat
NETosis markers in Patients before the walking test: circulating citrulinated histone H3 | Day 7
  The percentage of circulating citrulinated histone H3 will be measured on a SYSMEX automat
NETosis markers in Patients after the walking test: circulating citrulinated histone H3 | Day 7
  The percentage of circulating citrulinated histone H3 will be measured on a SYSMEX automat
Coagulation factors in Controls before the walking test: fibrinogen | Day 0
  Fibrinogen will be measured in g/L
Coagulation factors in Controls before the walking test | Day 0
  Coagulation factors XI, IX, VIII, VII, V, X and II will be measured in International Units
Coagulation factors in Controls after the walking test: fibrinogen | Day 0
  Fibrinogen will be measured in g/L
Coagulation factors in Controls after the walking test | Day 0
  Coagulation factors XI, IX, VIII, VII, V, X and II will be measured in International Units
Coagulation factors in Patients before the walking test: fibrinogen | Day 7
  Fibrinogen will be measured in g/L
Coagulation factors in Patients before the walking test | Day 7
  Coagulation factors XI, IX, VIII, VII, V, X and II will be measured in International Units
Coagulation factors in Patients after the walking test: fibrinogen | Day 7
  Fibrinogen will be measured in g/L
Coagulation factors in Patients after the walking test | Day 7
  Coagulation factors XI, IX, VIII, VII, V, X and II will be measured in International Units
Indicators of fibrinoformation in Controls before the walking test: circulating fibrin monomers | Day 0
  Circulating fibrin monomers will be measured in fibrinogen equivalent units
Indicators of fibrinoformation in Controls after the walking test: circulating fibrin monomers | Day 0
  Circulating fibrin monomers will be measured in fibrinogen equivalent units
Indicators of fibrinoformation in Controls before the walking test: circulating fibrin monomers | Day 7
  Circulating fibrin monomers will be measured in fibrinogen equivalent units
Indicators of fibrinoformation in Controls after the walking test: circulating fibrin monomers | Day 7
  Circulating fibrin monomers will be measured in fibrinogen equivalent units
Indicators of fibrinoformation in Patients before the walking test: circulating fibrin monomers | Day 0
  Circulating fibrin monomers will be measured in fibrinogen equivalent units
Indicators of fibrinoformation in Patients after the walking test: circulating fibrin monomers | Day 0
  Circulating fibrin monomers will be measured in fibrinogen equivalent units
Indicators of fibrinoformation in Patients before the walking test: circulating fibrin monomers | Day 7
  Circulating fibrin monomers will be measured in fibrinogen equivalent units
Indicators of fibrinoformation in Patients after the walking test: circulating fibrin monomers | Day 7
  Circulating fibrin monomers will be measured in fibrinogen equivalent units
Indicators of fibrinoformation in Controls before the walking test: D-dimers | Day 0
  D-dimers will be measured in DDUs
Indicators of fibrinoformation in Controls after the walking test: D-dimers | Day 0
  D-dimers will be measured in DDUs
Indicators of fibrinoformation in Patients before the walking test: D-dimers | Day 0
  D-dimers will be measured in DDUs
Indicators of fibrinoformation in Patients after the walking test: D-dimers | Day 0
  D-dimers will be measured in DDUs
Indicators of fibrinoformation in Controls before the walking test: D-dimers | Day 7
  D-dimers will be measured in DDUs
Indicators of fibrinoformation in Controls after the walking test: D-dimers | Day 7
  D-dimers will be measured in DDUs
Indicators of fibrinoformation in Patients before the walking test: D-dimers | Day 7
  D-dimers will be measured in DDUs
Indicators of fibrinoformation in Patients after the walking test: D-dimers | Day 7
  D-dimers will be measured in DDUs
Markers of fibrinolysis in Controls before the walking test : Euglobulin lysis time | Day 0
  Euglobulin lysis time will be measured in hours
Markers of fibrinolysis in Controls after the walking test : Euglobulin lysis time | Day 0
  Euglobulin lysis time will be measured in hours
Markers of fibrinolysis in Patients before the walking test : Euglobulin lysis time | Day 0
  Euglobulin lysis time will be measured in hours
Markers of fibrinolysis in Patients after the walking test : Euglobulin lysis time | Day 0
  Euglobulin lysis time will be measured in hours
Markers of fibrinolysis in Controls before the walking test : Euglobulin lysis time | Day 7
  Euglobulin lysis time will be measured in hours
Markers of fibrinolysis in Controls after the walking test : Euglobulin lysis time | Day 7
  Euglobulin lysis time will be measured in hours
Markers of fibrinolysis in Patients before the walking test : Euglobulin lysis time | Day 7
  Euglobulin lysis time will be measured in hours
Markers of fibrinolysis in Patients after the walking test : Euglobulin lysis time | Day 7
  Euglobulin lysis time will be measured in hours
Markers of Endothelial function in Controls before the walking test: Willebrand factor | Day 0
  Willebrand factor will be measured as a %
Markers of Endothelial function in Controls after the walking test: Willebrand factor | Day 0
  Willebrand factor will be measured as a %
Markers of Endothelial function in Patients before the walking test: Willebrand factor | Day 0
  Willebrand factor will be measured as a %
Markers of Endothelial function in Patients after the walking test: Willebrand factor | Day 0
  Willebrand factor will be measured as a %
Markers of Endothelial function in Controls before the walking test: Willebrand factor | Day 7
  Willebrand factor will be measured as a %
Markers of Endothelial function in Controls after the walking test: Willebrand factor | Day 7
  Willebrand factor will be measured as a %
Markers of Endothelial function in Patients before the walking test: Willebrand factor | Day 7
  Willebrand factor will be measured as a %
Markers of Endothelial function in Patients after the walking test: Willebrand factor | Day 7
  Willebrand factor will be measured as a%
Markers of Endothelial function in Controls before the walking test: ristocetin cofactor | Day 0
  Ristocetin cofactor will be measured as a %
Markers of Endothelial function in Controls after the walking test: ristocetin cofactor | Day 0
  Ristocetin cofactor will be measured as a %
Markers of Endothelial function in Patients before the walking test: ristocetin cofactor | Day 0
  Ristocetin cofactor will be measured as a %
Markers of Endothelial function in Patients after the walking test: ristocetin cofactor | Day 0
  Ristocetin cofactor will be measured as a %
Markers of Endothelial function in Controls before the walking test: ristocetin cofactor | Day 7
  Ristocetin cofactor will be measured as a %
Markers of Endothelial function in Controls after the walking test: ristocetin cofactor | Day 7
  Ristocetin cofactor will be measured as a %
Markers of Endothelial function in Patients before the walking test: ristocetin cofactor | Day 7
  Ristocetin cofactor will be measured as a %
Markers of Endothelial function in Patients after the walking test: ristocetin cofactor | Day 7
  Ristocetin cofactor will be measured as a %
Markers of Endothelial function in Controls before the walking test: ADAMTS-13 activity | Day 0
  ADAMTS-13 activity will be measured as a %
Markers of Endothelial function in Controls after the walking test: ADAMTS-13 activity | Day 0
  ADAMTS-13 activity will be measured as a %
Markers of Endothelial function in Patients before the walking test: ADAMTS-13 activity | Day 0
  ADAMTS-13 activity will be measured as a %
Markers of Endothelial function in Patients after the walking test: ADAMTS-13 activity | Day 0
  ADAMTS-13 activity will be measured as a %
Markers of Endothelial function in Controls before the walking test: ADAMTS-13 activity | Day 7
  ADAMTS-13 activity will be measured as a %
Markers of Endothelial function in Controls after the walking test: ADAMTS-13 activity | Day 7
  ADAMTS-13 activity will be measured as a %
Markers of Endothelial function in Patients before the walking test: ADAMTS-13 activity | Day 7
  ADAMTS-13 activity will be measured as a %
Markers of Endothelial function in Patients after the walking test: ADAMTS-13 activity | Day 7
  ADAMTS-13 activity will be measured as a %
Markers of Endothelial function in Controls before the walking test: soluble thrombomodulin | Day 0
  Soluble thrombomodulin will be measured as a %
Markers of Endothelial function in Controls after the walking test: soluble thrombomodulin | Day 0
  Soluble thrombomodulin will be measured as a %
Markers of Endothelial function in Patients before the walking test: soluble thrombomodulin | Day 0
  Soluble thrombomodulin will be measured as a %
Markers of Endothelial function in Patients after the walking test: soluble thrombomodulin | Day 0
  Soluble thrombomodulin will be measured as a %
Markers of Endothelial function in Controls before the walking test: soluble thrombomodulin | Day 7
  Soluble thrombomodulin will be measured as a %
Markers of Endothelial function in Controls after the walking test: soluble thrombomodulin | Day 7
  Soluble thrombomodulin will be measured as a %
Markers of Endothelial function in Patients before the walking test: soluble thrombomodulin | Day 7
  Soluble thrombomodulin will be measured as a %
Markers of Endothelial function in Patients after the walking test: soluble thrombomodulin | Day 7
  Soluble thrombomodulin will be measured as a %
Markers of Endothelial function in Controls before the walking test: soluble endothelial protein C receptor | Day 0
  Soluble endothelial protein C receptor will be measured as a %
Markers of Endothelial function in Controls after the walking test: soluble endothelial protein C receptor | Day 0
  Soluble endothelial protein C receptor will be measured as a %
Markers of Endothelial function in Patients before the walking test: soluble endothelial protein C receptor | Day 0
  Soluble endothelial protein C receptor will be measured as a %
Markers of Endothelial function in Patients after the walking test: soluble endothelial protein C receptor | Day 0
  Soluble endothelial protein C receptor will be measured as a %
Markers of Endothelial function in Controls before the walking test: soluble endothelial protein C receptor | Day 7
  Soluble endothelial protein C receptor will be measured as a %
Markers of Endothelial function in Controls after the walking test: soluble endothelial protein C receptor | Day 7
  Soluble endothelial protein C receptor will be measured as a %
Markers of Endothelial function in Patients before the walking test: soluble endothelial protein C receptor | Day 7
  Soluble thrombomodulin will be measured as a %
Markers of Endothelial function in Patients after the walking test: soluble endothelial protein C receptor | Day 7
  Soluble thrombomodulin will be measured as a %

OTHER OUTCOMES:
Age in Controls | Day 0
  Ages will be recorded in years
Sex in Controls | Day 0
  Sex will be recorded as Male/Female/Non-binary
Body mass index in Controls | Day 0
  Body mass index of controls will be recorded in units of kg/m²
Age in Patients | Day 0
  Ages will be recorded in years
Sex in Patients | Day 0
  Sex will be recorded as Male/Female/Non-binary
Body Mass Index in Patients | Day 0
  Body mass index of controls will be recorded in units of kg/m²

CONTACTS AND LOCATIONS:
Overall Officials: Antonia PEREZ MARTIN, Prof., Principal Investigator — Nîmes University Hospital; Stéphane FAURE, Principal Investigator — Nîmes University Hospital
Locations (1):
- CHU de Nîmes, Nîmes, Occitanie, France

REFERENCES:
- [Background] Gris JC, Guillotin F, Dos Santos TP, Chea M, Loubet P, Laureillard D, Sotto A, Muller L, Barbar SD, Roger C, Lefrant JY, Jung B, Klouche K, Mura T, Quere I, Perez-Martin A. Prognostic value of an automated thrombin generation assay in COVID-19 patients entering hospital: A multicentric, prospective observational study. Thromb Res. 2023 Feb;222:85-95. doi: 10.1016/j.thromres.2022.12.019. Epub 2023 Jan 2. PMID 36608393